CLINICAL TRIAL: NCT03207841
Title: Utilizing a Low-Carbohydrate/High-Protein Diet to Improve Metabolic Health in Individuals With Spinal Cord Injury
Brief Title: Low Carbohydrate/High Protein Diet to Improve Metabolic Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University (Other)
Responsible Party: Principal Investigator, Ceren Yarar-Fisher, Principal Investigator, Ohio State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: HHS-2016-ACL-NIDILRR-SI-0158
Record Dates: First submitted 2017-06-27; First posted 2017-07-05 (Actual); Last update posted 2023-03-27 (Actual); Status verified 2023-03

CONDITIONS: Spinal Cord; Metabolic Syndrome; Diabetes
Keywords: SCI; High Protein; Low Carbohydrate; Metabolic Health; Microbiome
MeSH Terms: conditions — Metabolic Syndrome; Diabetes Mellitus

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LC/HP group (Experimental): Intervention group will receive 8 weeks of LC/HP diet. The daily LC-HP dietary intervention will include ~30% total energy as protein (1.6 g/kg per day) with a carbohydrate-to-protein ratio <1.5 and fat intake set at ~30% of the total energy intake. Dietary fat sources will focus on monounsaturated and polyunsaturated fats, e.g., plant oils and nuts; dietary carbohydrate sources will emphasize whole grains, fruits, vegetables, and legumes; and dietary protein sources will include lean meats, fish, chicken, eggs, and nonfat dairy foods, e.g., fat-free milk and low-fat cheese, consistent with American Diabetes Association and Institute of Medicine guidelines. All LC-HP meals will be provided by UAB Center for Clinical and Translational Sciences (CCTS) Bionutrition Unit and delivered to participants' homes 3 times/week (a sample menu is included in Appendix J). Every delivery will include breakfast, lunch, dinner, and snacks for 2 to 3 days.
  Interventions: Other: LC/HP
- Control (No Intervention): Control group will not receive the experimental diet and will continue with their usual diets. Participants will complete three 24-hour food recalls (on 2 week days and one day in the weekend) three times (at weeks 1, 4 and 8) during the course of the study to gather dietary information including dietary intake and/or particular aspects of the diet. Participants will be asked to recall foods and beverages they consumed in the 24 hours prior to the interview. Three 24-hour food recalls appear optimal for estimating energy intake.

INTERVENTIONS:
Other: LC/HP — Intervention group will receive 8 weeks of LC/HP diet. The daily LC-HP dietary intervention will include ~30% total energy as protein (1.6 g/kg per day) with a carbohydrate-to-protein ratio <1.5 and fat intake set at ~30% of the total energy intake.
  Arms: LC/HP group

SUMMARY:
Individuals with spinal cord injury (SCI) are living to ages when metabolic disorders are highly prevalent. The combination of impaired glucose tolerance and insulin resistance can disrupt lipid metabolism and increase the risk of cardiovascular disease and diabetes, and contribute to an accelerated aging process in the SCI population. Feasible interventions to improve metabolic function in the chronic SCI are in great demand. Compared to pharmacologic therapies, dietary modification is a more cost-effective treatment option for reducing the risk of metabolic dysfunction that, surprisingly, has not been rigorously investigated in people with SCI. Therefore, in the present study the investigators will investigate the efficacy of an 8-week, eucaloric (a meal plan designed specifically to provide the exact amount of calories needed to maintain a given body weight) LC-HP dietary intervention for improving metabolic function, body composition, gut bacteria composition and quality of life in individuals with SCI and impaired glucose tolerance or type 2 diabetes. The investigators also aim to determine the association between changes in the composition of gut bacteria and improvements in metabolic function and the association between improvements in metabolic function and improvements in quality of life.

DETAILED DESCRIPTION:
Individuals with spinal cord injury (SCI) are living to ages when metabolic disorders are highly prevalent. Due to the loss of mobility and severe skeletal muscle atrophy in individuals with SCI, obesity, impaired glucose tolerance, and peripheral insulin resistance develop after injury . The combination of impaired glucose tolerance and insulin resistance can disrupt lipid metabolism and increase the risk of cardiovascular disease and diabetes, and contribute to an accelerated aging process in the SCI population. Because of these trends, the overall burden of health complications and their economic impact has increased for individuals with SCI, often leading to a progressive decrease in their long-term quality of life. Feasible interventions to improve metabolic function (i.e. the way the body processes proteins, carbohydrates, and fats in foods) in those with chronic SCI are in great demand. Given that metabolic disorders severely compromise health outcomes and important domains of quality of life, including participation in daily life and community living and employment outcomes, targeted strategies to combat these morbidities are of paramount importance. Compared to pharmacologic therapies, dietary modification is a more cost-effective treatment option for reducing the risk of metabolic dysfunction that, surprisingly, has not been rigorously investigated in people with SCI. Much like the general U.S. population, individuals with SCI consume far more fat and carbohydrate than recommended levels. High fat, high carbohydrate diets (western diet) have been associated with a higher prevalence of obesity and metabolic disease as well as negative adaptations in the diversity of gut bacteria (increased levels of harmful bacteria and reduced levels of beneficial bacteria) that usually precedes the development of diabetes or insulin resistance. Therefore, macronutrient (carbohydrate, protein, and fat) modification may be able to prevent or correct the impaired metabolic state in persons with SCI. Diets composed of relatively high protein and low carbohydrate have been shown to improve body composition (i.e., reduce body fat while maintaining lean tissue) and metabolic profiles (i.e., increase in insulin sensitivity and glucose tolerance) in diabetic, able bodied individuals who are obese or overweight. This improvement is thought to be due to protein's: (i) effect on the sensation of feeling full after eating food despite similar or lower energy intake; (ii) contribution to storage of fat-free mass; and (iii) insulin sensitizing effect.

The investigators' pilot work supports this hypothesis in that we showed that 8 weeks of a low carbohydrate/high-protein (LC-HP) diet significantly improved whole body insulin sensitivity (WBIS) and glucose tolerance and decreased the amount of intra-abdominal fat in six men with SCI and with either untreated type 2 diabetes or impaired glucose tolerance (pre-diabetes). In addition to significant improvements in metabolic health, our pilot work also successfully demonstrated the safety and feasibility of our approach. The lack of adverse effects and the improvement in glucose control and insulin sensitivity in our study participants with SCI prompted us to propose the current study involving both men and women in order to determine the effects of the dietary protocol to treat type 2 diabetes or impaired glucose tolerance in persons with chronic SCI. Thus, the investigators propose an investigation to determine if 8 weeks of an LC/HP dietary intervention induces the physiological adaptations necessary to improve metabolic function and body composition and alter the diversity of gut bacteria in a large cohort of individuals with SCI. The ultimate outcome of this project will be an effective diet program which can be easily and economically implemented at home as a non-pharmacological means of achieving blood glucose control for people with SCI and impaired glucose tolerance or untreated type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 18 and 65 years
* diagnosis of traumatic SCI at the cervical, thoracic, or lumbar level (C5-L2) classified as American Spinal Cord Injury Association Classification (AIS) A, B, C, or D
* Impaired glucose tolerance or untreated type 2 diabetes
* at least 3 years post-injury.

Exclusion Criteria:

* Pregnant women.
* Neurological (other than SCI), vascular and/or cardiac problems that may limit function and interfere with testing procedures
* Patients with evidence of renal insufficiency and liver disease by history, physical examination, and laboratory tests
* Patients with underlying pulmonary diseases

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2022-08-01 (Actual); Study Completion 2022-08-29 (Actual)

PRIMARY OUTCOMES:
Change in glucose tolerance | Week1 and Week 8
Change in insulin sensitivity | Week 1 and Week 8
Change in body mass index | Week 1 and Week 8
Change in gut bacterial composition | Week 1 and Week 8
Change in HDL, LDL, total cholesterol and triglycerides | Week 1 and Week 8

SECONDARY OUTCOMES:
Change in Spinal Cord Injury-Quality of Life (SCI-QOL) Score | Week 1 and Week 8

CONTACTS AND LOCATIONS:
Locations (1):
- UAB, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Li J, Gower B, McLain A, Yarar-Fisher C. Effects of a low-carbohydrate/high-protein diet on metabolic health in individuals with chronic spinal cord injury: An exploratory analysis of results from a randomized controlled trial. Physiol Rep. 2022 Nov;10(22):e15501. doi: 10.14814/phy2.15501. PMID 36411989
- [Derived] Li J, Morrow C, McLain A, Womack ED, Yarar-Fisher C. Effects of a Low-Carbohydrate, High-Protein Diet on Gut Microbiome Composition in Insulin-Resistant Individuals With Chronic Spinal Cord Injury: Preliminary Results From a Randomized Controlled Trial. Arch Phys Med Rehabil. 2022 Jul;103(7):1269-1278. doi: 10.1016/j.apmr.2022.03.014. Epub 2022 Apr 10. PMID 35417758
- [Derived] Yarar-Fisher C, Li J, McLain A, Gower B, Oster R, Morrow C. Utilizing a low-carbohydrate/high-protein diet to improve metabolic health in individuals with spinal cord injury (DISH): study protocol for a randomized controlled trial. Trials. 2019 Jul 30;20(1):466. doi: 10.1186/s13063-019-3520-3. PMID 31362773